CLINICAL TRIAL: NCT05013749
Title: Hysterectomy Vs Partial Myometrial Resection for Placenta Accreta Spectrum (PAS). A Feasibility Study of a Randomized Controlled Clinical Experiment (RCT-PAS)
Brief Title: Histerectomy Vs Partial Myometrial Resection for Placenta Accreta Spectrum
Acronym: RCT-PAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Clinica Valle del Lili (Other)
Responsible Party: Principal Investigator, Albaro Nieto, Gynecologist and Obstetrician, Fundacion Clinica Valle del Lili
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1751
Record Dates: First submitted 2021-07-22; First posted 2021-08-19 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Placenta Accreta
Keywords: Placenta accreta; Resective reconstructive treatment; Hysterectomy
MeSH Terms: conditions — Placenta Accreta | interventions — Hysterectomy

STUDY DESIGN:
Intervention Model Description: Eligible women will receive complete information about the study. If they agree to participate in it, they will sign the informed consent for both interventions: hysterectomy and partial myometrial resection. The final modality of intervention will be decided at randomization prior to the start of the surgical procedure.
  If the diagnosis of PAS is confirmed by observing the clinical criteria endorsed by the International Federation of Gynecology and Obstetrics (FIGO), the patient's participation in the study is confirmed and the surgical procedure defined by randomization is continued, that is, one of the two arms of the study: Primary hysterectomy or Partial myometrial resection.
Masking Description: This is an open-label study as it is not possible to conceal the surgical procedure for each arm from the operator (Treating Physician) or from the participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hysterectomy (Active Comparator): Hysterectomy: An incision will be made above the level of the placenta, delivering the newborn. Uterotonics will be administered, and spontaneous delivery of the placenta will be awaited using gentle traction. The absence of spontaneous separation of the placenta will confirm the diagnosis of PAS, the patient will undergo to hysterectomy. The complete removal of the uterus will be attempted, including the cervix, the duration of the intervention and intraoperative blood loss will be recorded, as well as the damage to organs neighboring the uterus. In this arm of the study, to hysterectomy will be performed in 100% of patients
  Interventions: Procedure: Hysterectomy
- Partial myometrial resection (Active Comparator): Partial myometrial resection: The technique described by Palacios-Jaraquemada et al5. will be followed. Briefly, the uterus will be dissected to free it from the posterior wall of the bladder to the cervix. The vesicouterine vessels will be ligated and the parametrial space will be visualized. The hysterotomy will be performed in the upper segment, immediately above the area of invasion of the myometrium. The entire invaded myometrium and the entire placenta will be removed. The uterus will repair itself in one or two layers. Intrauterine balloon tamponade will be used if indicated.
  Interventions: Procedure: Partial Myometrial Resection

INTERVENTIONS:
Procedure: Hysterectomy — Hysterectomy: An incision will be made above the level of the placenta, delivering the newborn. Uterotonics will be administered, and spontaneous delivery of the placenta will be awaited using gentle traction. The absence of spontaneous separation of the placenta will confirm the diagnosis of PAS, the patient will undergo to hysterectomy. The complete removal of the uterus will be attempted, including the cervix, the duration of the intervention and intraoperative blood loss will be recorded, as well as the damage to organs neighboring the uterus. In this arm of the study, to hysterectomy will be performed in 100% of patients
  Arms: Hysterectomy
Procedure: Partial Myometrial Resection — Partial myometrial resection: The technique described by Palacios-Jaraquemada et al5. will be followed. Briefly, the uterus will be dissected to free it from the posterior wall of the bladder to the cervix. The vesico-uterine vessels will be ligated and the parametrial space will be visualized. The hysterotomy will be performed in the upper segment, immediately above the area of invasion of the myometrium. The entire invaded myometrium and the entire placenta will be removed. The uterus will repair itself in one or two layers. Intrauterine balloon tamponade will be used if indicated.
  Arms: Partial myometrial resection

SUMMARY:
Currently, Placenta Accreta Spectrum (PAS) has two treatment options: hysterectomy (completely removing the uterus) and partial myometrial resection (resecting the part of the uterus affected by this pathology).

The present study is a feasibility study of a multicenter, randomized controlled clinical trial to be carried out in 3 health institutions. Patients who meet the inclusion criteria, after signing the informed consent, will be taken to the surgical procedure and before the start of the procedure they will be randomized to one of the two interventions, hysterectomy or partial myometrial resection, intra-surgical clinical outcomes will be explored and a follow-up will be carried out during the immediate post-surgical period (72 hours), in 7 to 12 days and at 42 days postpartum.

A sample size of 60 patients is estimated among the 3 health institutions, with an approximate duration of the study of 24 months.

DETAILED DESCRIPTION:
Placenta accreta spectrum is a serious condition associated with significant maternal morbidity and even mortality. The recommended treatment is hysterectomy. An alternative is 1-step conservative surgery, which involves the en bloc resection of the myometrium affected by placenta accreta spectrum along with the placenta, followed by uterine reconstruction. Currently, there are no studies comparing the 2 techniques in the setting of a randomized controlled trial.

We performed a prospectively registered multicenter randomized controlled trial comparing hysterectomy with 1-step conservative surgery. The aim was to collect feasibility and clinical outcomes of the 2 techniques in women assigned to hysterectomy or 1step conservative surgery. In addition to assessing participants' willingness to be randomized, we also collected data on intraoperative blood loss, transfusion requirement, serious adverse event, and other clinical outcomes.

Sixty women with strong antenatal suspicion of placenta accreta spectrum were assigned randomly to either hysterectomy (n=31) or 1-step conservative surgery (n=29).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women over 18 years of age.
* History of previous cesarean section and anterior placenta previa
* Patients with prenatal diagnosis by ultrasound or MRI of PAS, regardless of the suspected degree of severity of the disease.
* Requirement for surgical management of placental accreta on a scheduled basis.
* Patients without active vaginal bleeding in the period immediately before surgery (Patients entering the operating room without active bleeding).

Exclusion Criteria:

* Women without previous living children.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albaro Nieto-Calvache, MD, Principal Investigator — Fundacion Clinica Valle del Lili
Locations (1):
- Fundación Valle del Lili, Cali, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silver RM, Landon MB, Rouse DJ, Leveno KJ, Spong CY, Thom EA, Moawad AH, Caritis SN, Harper M, Wapner RJ, Sorokin Y, Miodovnik M, Carpenter M, Peaceman AM, O'Sullivan MJ, Sibai B, Langer O, Thorp JM, Ramin SM, Mercer BM; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Maternal morbidity associated with multiple repeat cesarean deliveries. Obstet Gynecol. 2006 Jun;107(6):1226-32. doi: 10.1097/01.AOG.0000219750.79480.84. PMID 16738145
- [Background] D'Antonio F, Iacovella C, Bhide A. Prenatal identification of invasive placentation using ultrasound: systematic review and meta-analysis. Ultrasound Obstet Gynecol. 2013 Nov;42(5):509-17. doi: 10.1002/uog.13194. Epub 2013 Oct 2. PMID 23943408
- [Background] Jauniaux E, Bhide A. Prenatal ultrasound diagnosis and outcome of placenta previa accreta after cesarean delivery: a systematic review and meta-analysis. Am J Obstet Gynecol. 2017 Jul;217(1):27-36. doi: 10.1016/j.ajog.2017.02.050. Epub 2017 Mar 6. PMID 28268196
- [Background] Fitzpatrick KE, Sellers S, Spark P, Kurinczuk JJ, Brocklehurst P, Knight M. The management and outcomes of placenta accreta, increta, and percreta in the UK: a population-based descriptive study. BJOG. 2014 Jan;121(1):62-70; discussion 70-1. doi: 10.1111/1471-0528.12405. Epub 2013 Aug 7. PMID 23924326
- [Background] Nieto AJ, Echavarria MP, Carvajal JA, Messa A, Burgos JM, Ordonez C, Benavidez JP, Mejia M, Lopez L, Fernandez PA, Escobar MF. Placenta accreta: importance of a multidisciplinary approach in the Colombian hospital setting. J Matern Fetal Neonatal Med. 2020 Apr;33(8):1321-1329. doi: 10.1080/14767058.2018.1517328. Epub 2018 Sep 25. PMID 30153754
- [Background] Collins SL, Alemdar B, van Beekhuizen HJ, Bertholdt C, Braun T, Calda P, Delorme P, Duvekot JJ, Gronbeck L, Kayem G, Langhoff-Roos J, Marcellin L, Martinelli P, Morel O, Mhallem M, Morlando M, Noergaard LN, Nonnenmacher A, Pateisky P, Petit P, Rijken MJ, Ropacka-Lesiak M, Schlembach D, Sentilhes L, Stefanovic V, Strindfors G, Tutschek B, Vangen S, Weichert A, Weizsacker K, Chantraine F; International Society for Abnormally Invasive Placenta (IS-AIP). Evidence-based guidelines for the management of abnormally invasive placenta: recommendations from the International Society for Abnormally Invasive Placenta. Am J Obstet Gynecol. 2019 Jun;220(6):511-526. doi: 10.1016/j.ajog.2019.02.054. Epub 2019 Mar 5. PMID 30849356
- [Background] Palacios-Jaraquemada JM, Fiorillo A, Hamer J, Martinez M, Bruno C. Placenta accreta spectrum: a hysterectomy can be prevented in almost 80% of cases using a resective-reconstructive technique. J Matern Fetal Neonatal Med. 2022 Jan;35(2):275-282. doi: 10.1080/14767058.2020.1716715. Epub 2020 Jan 26. PMID 31984808
- [Background] Allen L, Jauniaux E, Hobson S, Papillon-Smith J, Belfort MA; FIGO Placenta Accreta Diagnosis and Management Expert Consensus Panel. FIGO consensus guidelines on placenta accreta spectrum disorders: Nonconservative surgical management. Int J Gynaecol Obstet. 2018 Mar;140(3):281-290. doi: 10.1002/ijgo.12409. No abstract available. PMID 29405317
- [Background] Sentilhes L, Kayem G, Chandraharan E, Palacios-Jaraquemada J, Jauniaux E; FIGO Placenta Accreta Diagnosis and Management Expert Consensus Panel. FIGO consensus guidelines on placenta accreta spectrum disorders: Conservative management. Int J Gynaecol Obstet. 2018 Mar;140(3):291-298. doi: 10.1002/ijgo.12410. No abstract available. PMID 29405320
- [Background] Nieto-Calvache AJ, Lopez-Giron MC, Messa-Bryon A, Ceballos-Posada ML, Duque-Galan M, Rios-Posada JG, Plazas-Cordoba LA, Chancy-Castano MM. Urinary tract injuries during treatment of patients with morbidly adherent placenta. J Matern Fetal Neonatal Med. 2021 Oct;34(19):3140-3146. doi: 10.1080/14767058.2019.1678135. Epub 2019 Oct 21. PMID 31631730
- [Background] Nieto-Calvache AJ, Vergara-Galliadi LM, Rodriguez F, Ordonez CA, Garcia AF, Lopez MC, Manzano R, Velasquez J, Carbonell JP, Bryon AM, Echavarria MP, Escobar MF, Carvajal J, Benavides-Calvache JP, Burgos JM. A multidisciplinary approach and implementation of a specialized hemorrhage control team improves outcomes for placenta accreta spectrum. J Trauma Acute Care Surg. 2021 May 1;90(5):807-816. doi: 10.1097/TA.0000000000003090. PMID 33496549
- [Background] Nieto-Calvache AJ, Lopez-Giron MC, Quintero-Santacruz M, Bryon AM, Burgos-Luna JM, Echavarria-David MP, Lopez L, Macia-Mejia C, Benavides-Calvache JP. A systematic multidisciplinary initiative may reduce the need for blood products in patients with abnormally invasive placenta. J Matern Fetal Neonatal Med. 2022 Feb;35(4):738-744. doi: 10.1080/14767058.2020.1731460. Epub 2020 Feb 23. PMID 32089029
- [Background] Nieto-Calvache AJ, Zambrano MA, Herrera NA, Usma A, Bryon AM, Benavides Calvache JP, Lopez L, Mejia M, Palacios-Jaraquemada JM. Resective-reconstructive treatment of abnormally invasive placenta: Inter Institutional Collaboration by telemedicine (eHealth). J Matern Fetal Neonatal Med. 2021 Mar;34(5):765-773. doi: 10.1080/14767058.2019.1615877. Epub 2019 May 27. PMID 31057039
- [Background] Teixidor Vinas M, Belli AM, Arulkumaran S, Chandraharan E. Prevention of postpartum hemorrhage and hysterectomy in patients with morbidly adherent placenta: a cohort study comparing outcomes before and after introduction of the Triple-P procedure. Ultrasound Obstet Gynecol. 2015 Sep;46(3):350-5. doi: 10.1002/uog.14728. PMID 25402727
- [Background] Pinas Carrillo A, Chandraharan E. Placenta accreta spectrum: Risk factors, diagnosis and management with special reference to the Triple P procedure. Womens Health (Lond). 2019 Jan-Dec;15:1745506519878081. doi: 10.1177/1745506519878081. PMID 31578123
- [Background] Jauniaux E, Ayres-de-Campos D, Langhoff-Roos J, Fox KA, Collins S; FIGO Placenta Accreta Diagnosis and Management Expert Consensus Panel. FIGO classification for the clinical diagnosis of placenta accreta spectrum disorders. Int J Gynaecol Obstet. 2019 Jul;146(1):20-24. doi: 10.1002/ijgo.12761. PMID 31173360
- [Background] Jauniaux E, Bhide A, Kennedy A, Woodward P, Hubinont C, Collins S; FIGO Placenta Accreta Diagnosis and Management Expert Consensus Panel. FIGO consensus guidelines on placenta accreta spectrum disorders: Prenatal diagnosis and screening. Int J Gynaecol Obstet. 2018 Mar;140(3):274-280. doi: 10.1002/ijgo.12408. No abstract available. PMID 29405319
- [Background] Jha P, Poder L, Bourgioti C, Bharwani N, Lewis S, Kamath A, Nougaret S, Soyer P, Weston M, Castillo RP, Kido A, Forstner R, Masselli G. Society of Abdominal Radiology (SAR) and European Society of Urogenital Radiology (ESUR) joint consensus statement for MR imaging of placenta accreta spectrum disorders. Eur Radiol. 2020 May;30(5):2604-2615. doi: 10.1007/s00330-019-06617-7. Epub 2020 Feb 10. PMID 32040730
- [Derived] Nieto-Calvache AJ, Aryananda RA, Palacios-Jaraquemada JM, Cininta N, Grace A, Benavides-Calvache JP, Campos CI, Messa-Bryon A, Vallecilla L, Sarria D, Galindo JS, Galindo-Velasco V, Rivera-Torres LF, Burgos-Luna JM, Bhide A. One-step conservative surgery vs hysterectomy for placenta accreta spectrum: a feasibility randomized controlled trial. Am J Obstet Gynecol MFM. 2024 Jun;6(6):101333. doi: 10.1016/j.ajogmf.2024.101333. Epub 2024 Mar 6. PMID 38458362

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hysterectomy | Partial Myometrial Resection
Started | 31 | 29
Participants That Received a Different Intervention Than They Were Originally Randomized to | 7 | 9
Completed | 24 | 18
Not Completed | 7 | 11
Not completed — Patients without signs of PAS in the intraoperative staging. US false positive | 7 | 2
Not completed — Did not meet the requirements for OSCS after intraoperative staging. | 0 | 9

BASELINE CHARACTERISTICS:
Groups:
- Hysterectomy: An incision will be made above the level of the placenta, delivering the newborn. Uterotonics will be administered, and spontaneous delivery of the placenta will be awaited using gentle traction. The absence of spontaneous separation of the placenta will confirm the diagnosis of PAS, the patient will undergo to hysterectomy. The complete removal of the uterus will be attempted, including the cervix, the duration of the intervention and intraoperative blood loss will be recorded, as well as the damage to organs neighboring the uterus. In this arm of the study, to hysterectomy will be performed in 100% of patients
- Partial Myometrial Resection: The technique described by Palacios-Jaraquemada et al5. will be followed. Briefly, the uterus will be dissected to free it from the posterior wall of the bladder to the cervix. The vesicouterine vessels will be ligated and the parametrial space will be visualized. The hysterotomy will be performed in the upper segment, immediately above the area of invasion of the myometrium. The entire invaded myometrium and the entire placenta will be removed. The uterus will repair itself in one or two layers. Intrauterine balloon tamponade will be used if indicated.
- Total: Total of all reporting groups
Arm/Group | Hysterectomy | Partial Myometrial Resection | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Customized [Mean (Standard Deviation); unit: years]
  Maternal age (years) | 33.13 (4.26) | 33.45 (4.56) | 33.28 (4.38)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 31 | 29 | 60
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body mass index [Number; unit: kg/m^2] — Units used to assess Body mass index kg/m^2
  kg/m^2
    18-24 | 10 | 8 | 18
    25-29 | 13 | 12 | 25
    ≥30 | 8 | 9 | 17
Number of previous pregnancies [Number; unit: number of previous pregnancies]
  1 | 9 | 7 | 16
  2 | 16 | 8 | 24
  ≥3 | 6 | 14 | 20
Number of previous cesarean sections [Count of Participants; unit: Participants]
  1 | 18 | 14 | 32
  2 | 13 | 13 | 26
  ≥3 | 0 | 2 | 2
Number of previous dilatation curettage [Count of Participants; unit: Participants]
  0 | 24 | 21 | 45
  1 | 7 | 5 | 12
  ≥2 | 0 | 3 | 3
Gestational age at the time of diagnosis of PAS [Median (Inter-Quartile Range); unit: weeks] | 33.10 [31.50 to 34.70] | 31.00 [26.20 to 33.00] | 32.75 [30.00 to 34.10]
Diagnostic method of PAS [Count of Participants; unit: Participants]
  Ultrasound | 25 | 21 | 46
  Ultrasound and Magnetic Resonance | 6 | 8 | 14
Antepartum vaginal bleeding [Count of Participants; unit: Participants] | 1 | 0 | 1
Comorbidity [Number; unit: participants]
  Hypertensive disorder | 1 | 1 | 2
  Gestational diabetes | 0 | 1 | 1
Gestational age at birth [Median (Inter-Quartile Range); unit: weeks] | 35.00 [34.00 to 36.00] | 35.00 [34.00 to 36.00] | 35.00 [34.00 to 36.00]

OUTCOME MEASURES:

1. Primary Outcome: Feasibility: Proportion of Eligible Patients Who Agree to Participate in the Study.
Description: Number of patients who agree to participate, out of the total number of eligible patients
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Patients: Potential participants needed to have risk factors (placenta previa in the current pregnancy with at least one prior cesarean delivery) and suspected PAS according to ultrasound. Patients aged <18 years and those with active vaginal bleeding, no placenta previa, and no previous live children were excluded.
Arm/Group | Eligible Patients
Number analyzed (Participants) | 64
Participants | 60

2. Primary Outcome: Screening Failure Percentage
Description: Percentage of patients who entered the study but did not present macroscopic findings of placenta accreta spectrum during laparotomy.
Time Frame: During surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Hysterectomy | Partial Myometrial Resection
Number analyzed (Participants) | 31 | 29
Participants | 7 | 2

3. Primary Outcome: Percentage of Patients With Crossover Between Assigned Study Arms.
Description: All patients had been randomized before surgery to a certain procedure; however, after performing intraoperative staging, it was identified that some women did not have signs of PAS (7 patients with false positive prenatal diagnosis, randomized to hysterectomy), so they were managed with OSCS, and that some women did not meet the criteria to perform OSCS (9 patients randomized to OSCS), so they were managed with hysterectomy;
Time Frame: During surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Hysterectomy | Partial Myometrial Resection
Number analyzed (Participants) | 31 | 29
Participants | 7 | 9

4. Primary Outcome: Number of Participants Who Completed the Follow-up Evaluation.
Description: Number of participants who completed follow-up at 42 days postpartum
Time Frame: 42 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Hysterectomy | Partial Myometrial Resection
Number analyzed (Participants) | 31 | 29
Participants | 31 | 29

5. Secondary Outcome: Maternal Death
Description: Number of maternal deaths during the study period
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Hysterectomy | Partial Myometrial Resection
Number analyzed (Participants) | 31 | 29
Participants | 0 | 0

6. Secondary Outcome: Intra-surgical Bleeding Volume
Description: Surgical bleeding calculated in milliliters
Time Frame: During surgery
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Hysterectomy | Partial Myometrial Resection
Number analyzed (Participants) | 31 | 29
mL | 1500 [1122 to 2753] | 1740 [1010 to 2410]

7. Secondary Outcome: Blood Component Transfusion Requirement
Description: If during hospitalization the patient required transfusion of some type of blood component
Time Frame: Up to 42 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Hysterectomy | Partial Myometrial Resection
Number analyzed (Participants) | 31 | 29
Participants | 19 | 17

8. Secondary Outcome: Median Transfusion of Red Blood Cell Units (RBCU)
Description: Median number of units of red blood cells transfused
Time Frame: Up to 42 days postpartum
Measure: Median (Inter-Quartile Range); unit: Number of RBCU
Arm/Group | Hysterectomy | Partial Myometrial Resection
Number analyzed (Participants) | 31 | 29
Number of RBCU | 3 [2.5 to 4] | 2 [1 to 4]

9. Secondary Outcome: Number of Patients Who Met at Least 1 Near Miss Criterion
Description: Situation or indicator that almost led to a serious adverse event but did not actually result in harm. For this study, the event was cardiac arrest with successful resuscitation.
Time Frame: Up to 42 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Hysterectomy | Partial Myometrial Resection
Number analyzed (Participants) | 31 | 29
Participants | 1 | 0

10. Secondary Outcome: Number of Patients Who Had Bladder Injuries
Description: Number of patients who had intraoperative bladder injuries.
Time Frame: Up to 42 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Hysterectomy | Partial Myometrial Resection
Number analyzed (Participants) | 31 | 29
Participants | 2 | 1

11. Secondary Outcome: Number of Patients Who Need Surgical Reoperation.
Description: Number of patients who need surgical reoperation after index surgery
Time Frame: Up to 42 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Hysterectomy | Partial Myometrial Resection
Number analyzed (Participants) | 31 | 29
Participants | 1 | 1

12. Secondary Outcome: Number of Patients Who Were Admitted to the Intensive Care Unit.
Description: Number of patients that required management in the Intensive Care Unit
Time Frame: Up to 42 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Hysterectomy | Partial Myometrial Resection
Number analyzed (Participants) | 31 | 29
Participants | 4 | 3

13. Secondary Outcome: Number of Days of Postoperative Hospital Stay.
Description: Number of days of hospital stay after index surgery
Time Frame: Up to 42 days postpartum
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Hysterectomy | Partial Myometrial Resection
Number analyzed (Participants) | 31 | 29
Days | 4 [3.5 to 5] | 5 [3 to 6]

ADVERSE EVENTS:
Time Frame: Follow up to 42 days (6 weeks) postpartum.
Description: Five of the 8 women with adverse events were randomized to OSCS, but in 4 of them intraoperative staging led to an immediate crossover to hysterectomy, and OSCS was not attempted.
Arm/Group | Hysterectomy | Partial Myometrial Resection
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/27
Serious Adverse Events (participants affected / at risk) | 3/33 | 5/27
Other Adverse Events (participants affected / at risk) | 0/33 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hysterectomy (N=33) | Partial Myometrial Resection (N=27)
Adverse event (Surgical and medical procedures) | 3 | 5 — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term. Bleeding >2.5 L or other situation that prolonged hospitalization, motivated reoperation or rehospitalization, or put life at risk

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT05013749/Prot_SAP_002.pdf
  • Informed Consent Form (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT05013749/ICF_001.pdf